CLINICAL TRIAL: NCT00933998
Title: Restoration of Cutaneous Sensorum in Patients With Diabetic Peripheral Neuropathy (DPN) Via Metanx®
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carolina Musculoskeletal Institute (Other)
Collaborators: Pamlab, L.L.C. (Industry); Baylor University (Other)
Responsible Party: Principal Investigator, Mackie J. Walker, Jr., DPM, Medical Director, Podiatry Division, Carolina Musculoskeletal Institute
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMI-01
Record Dates: First submitted 2009-07-07; First posted 2009-07-08 (Estimated); Last update posted 2014-01-29 (Estimated); Status verified 2014-01

CONDITIONS: Diabetic Peripheral Neuropathy
Keywords: DPN
MeSH Terms: interventions — metanx; 5-methyltetrahydrofolate; mecobalamin; Pyridoxal Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Metanx (Experimental): Metanx bid for 2 weeks then daily. Compare to non treated patient population
  Interventions: Other: Metanx® (Oral L-methylfolate, Methylcobalamin and Pyridoxal 5'-phosphate)

INTERVENTIONS:
Other: Metanx® (Oral L-methylfolate, Methylcobalamin and Pyridoxal 5'-phosphate) — One pill twice a day for 2 weeks. Then one pill a day until 12 month study is up.
  Other Names: Metanx

SUMMARY:
The purpose of this research study is to determine if Metanx improves sensory neuropathy in persons with Type 2 diabetes. Metanx is a medical food available with a prescription from a physician. It consists of L-methylfolate, Pyridoxal 5'-phosphate, and Methylcobalamin, which are the active forms of folate, vitamin B6, and vitamin B12, respectively. Subjects will be assigned to receive Metanx for 12 months. Baseline quantitative sensory testing will be done before the patient receives Metanx. Additional quantitative sensory testing will be done at 6 and 12 months to evaluate.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive diabetic patients entering the office (private practice)
* Subjective symptoms of numbness, burning, paresthesia, etc.
* Failed Monofilament of at least two points on each foot
* Abnormal PSSD study
* Willing to participate in protocols or study

  * Taking one Metanx tablet bid for 2 weeks then one Metanx tablet daily
  * Keep scheduled appointments for follow up studies
  * Report any other medical interventions, studies, or medication changes
  * Report any problems of medical or psycho-social matters to investigators
  * HgbA1c NOT monitored or specific value required for participation

Exclusion Criteria:

* History of back problems (Surgery or ECSI) or other large fiber neuropathies
* History of chemotherapy
* History of chemical exposure

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-06; Primary Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Epidermal Nerve Density Count | 2 years
  Measure increase or decrease in ENFD count after 12 months of Metanx therapy in patients with diabetic peripheral neuropathy

CONTACTS AND LOCATIONS:
Locations (1):
- Carolina Musculoskeletal Institute, Aiken, South Carolina, United States